CLINICAL TRIAL: NCT06342908
Title: A Pilot Study to Evaluate the Safety and Feasibility of Neoantigen-Targeted Dendritic Cell Vaccination in Diffuse Hemispheric Glioma, H3 G34-Mutant
Brief Title: A Vaccine (Neoantigen-Targeted ppDC) for the Treatment of H3 G34-mutant Diffuse Hemispheric Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-001700; NCI-2024-00210 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-03-06; First posted 2024-04-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Hemispheric Glioma, H3 G34-Mutant
MeSH Terms: interventions — Specimen Handling; Leukapheresis; Magnetic Resonance Spectroscopy; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PpDC vaccine, Poly ICLC) (Experimental): Patients undergo leukapheresis 10 days prior to first injection. Patients then receive ppDC ID with poly ICLC IM in both arms Q2W for total 3 doses and then every 6 months for up to 3 doses. Patients undergo MRI throughout the trial. Patients also undergo blood sample collection throughout the trial in addition to stool sample collection during screening and on the trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Dendritic Cell Therapy; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Drug: Poly ICLC

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Dendritic Cell Therapy — Given PpDC vaccine ID
  Other Names: Dendritic Cell Vaccine Therapy
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Poly ICLC — Given IM
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid

SUMMARY:
This phase I trial tests the safety and side effects, and best dose of a vaccine (neoantigen-target ppDC) in treating patients with H3 G34-mutant diffuse hemispheric glioma. Vaccines made from the patient's own white blood cells and peptide-pulsed dendritic cells may help the body build an effective immune response to kill tumor cells. Giving neoantigen-targeted ppDC may be safe, tolerable and/or effective in treating patients with diffuse hemispheric glioma with a H3 G34 mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and feasibility of neoantigen-targeted ppDC in adult patients with diffuse hemispheric glioma (DHG).

SECONDARY OBJECTIVES:

I. To evaluate the immunogenicity of neoantigen-targeted ppDC in adult patients with DHG.

II. To determine whether neoantigen-targeted ppDC facilitates systemic T cell-mediated adaptive immune activation in DHG patients.

III. To determine whether neoantigen-targeted ppDC facilitates a target-specific anti-tumor T cell expansion in DHG patients.

IV. To determine whether pro-inflammatory phenotypic changes in systemic immune cell populations are detected in peripheral blood in response to neoantigen-targeted ppDC vaccination in DHG patients.

EXPLORATORY OBJECTIVES:

I. To estimate the potential efficacy of neoantigen-targeted ppDC in DHG patients.

II. To correlate physiologic and metabolic magnetic resonance imaging (MRI) with systemic immunologic response after neoantigen-targeted ppDC in DHG patients.

III. To isolate and sequence immunodominant anti-tumor T cell T-cell receptor (TCRs) stimulated by neoantigen-targeted ppDC in DHG patients.

IV. To explore whether study participants demonstrating immune-reactive responses to neoantigen-targeted ppDC harbor significantly different gastrointestinal microbiota profiles in comparison to unresponsive participants.

OUTLINE:

Patients undergo leukapheresis 10 days prior to first injection. Patients then receive ppDC intradermally (ID) with poly ICLC intramuscularly (IM) in both arms every 2 weeks (Q2W) for total 3 doses and then every 6 months for up to 3 doses. Patients undergo magnetic resonance imaging (MRI) throughout the trial. Patients also undergo blood sample collection throughout the trial in addition to stool sample collection during screening and on the trial.

After completion of study treatment, patients are followed up at 30 and 120 days and then up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18 and 50 years with pathologically-confirmed diagnosis of (or pathology re-review consistent with) DHG will be enrolled in this study
* A female participant who has childbearing potential must have negative urine or serum pregnancy test 72 hours prior to the first dose and be willing to use adequate method of contraception for course of study and 120 days after last dose
* The participant (or legally acceptable representative if applicable) provides informed consent (and written assent from minors) for the trial
* An interval of the following durations prior to enrollment:

  * At least 28 days from prior surgical resection
  * At least 14 days from prior stereotactic biopsy
* Have clinical pathology results, commercial targeted exome sequencing results, or sufficient archival tumor tissue to confirm DHG following registration. The following amount of tissue is preferred: 25-50 mg flash frozen tissue block. Formalin-fixed, paraffin embedded (FFPE) tissue block or 10 FFPE unstained slides (5µm thick) is acceptable at the discretion of the Sponsor-Investigator
* Have a Karnofsky performance status (KPS) ≥ 70
* Absolute neutrophil count (ANC) ≥ 1500/uL (specimens must be collected within 14 days prior to the start of study treatment)
* Platelets ≥ 100 000/µL (specimens must be collected within 14 days prior to the start of study treatment)
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (specimens must be collected within 14 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 week
* Creatinine or measured or calculated b creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 × ULN or ≥ 30 mL/min for participant with creatinine levels > 1.5 × institutional ULN (specimens must be collected within 14 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard.
* Total bilirubin ≤ 1.5 ×ULN or direct bilirubin ≤ ULN for participants with total bilirubin levels >1.5 × ULN (specimens must be collected within 14 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases) (specimens must be collected within 14 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (specimens must be collected within 14 days prior to the start of study treatment)

Exclusion Criteria:

* Age > 50 years or < 18 years
* Have had more than 1 separately-treated recurrences of the index tumor
* A woman of child-bearing potential who has a positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to enrollment. Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to ≤ grade 1 or baseline. Participants with ≤ grade 2 neuropathy may be eligible
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic corticosteroid therapy (dosing exceeding 1 mg/kg/day of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] is detected) infection. Note: no testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a known history of active tuberculosis (Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Kidney dysfunction precluding administration of gadolinium-based contrast
* Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-03-08 (Estimated); Study Completion 2028-01-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of regimen-limiting toxicities | Up to 120 days after last dose
  Will be graded in severity according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE, v 5.0) guidelines, monitoring for 30 days following each dose for adverse event recording, and for 120 days following each dose for serious adverse event recording.

SECONDARY OUTCOMES:
Significant increase in gamma-interferon (IFN) gene expression signature | Up to 4 years
  Peripheral blood mononuclear cells (PBMCs) will be evaluated by ribonucleic acid sequence for significant increase in gamma-interferon (IFN) gene expression signature, comparing baseline PBMCs with PBMCs obtained after each dose phase of peptide-pulsed dendritic cells (ppDC).
Significant clonal T cell expansion | Up to 4 years
  PBMCs obtained before and after each ppDC dose phase will be analyzed for significant clonal T cell expansion by bulk V beta-T cell receptor (TCR) sequencing.
Targets of clonal cytotoxic T cell expansion | Up to 4 years
  The targets of clonal cytotoxic T cell expansion in PBMCs in response to ppDC assessed by using target-specific major histocompatibility complex (MHC) oligomers binding assays.
Pro-inflammatory phenotypic changes in immune cell populations | Up to 4 years
  The pro-inflammatory phenotypic changes in immune cell populations in response to ppDC assessed by cellular indexing of transcriptomes, epitopes-sequencing and a multi-color fluorescence-activated cell sorting panel.
Changes in immune cell subset expansion and contraction in T cell and myeloid-derived cell populations | Up to 4 years
  The changes in immune cell subset expansion and contraction in T cell and myeloid-derived cell populations in response to ppDC assessed by cellular indexing of transcriptomes and epitopes-sequencing and a multi-color fluorescence-activated cell sorting panel.
Changes of immune cell markers profile in T cell and myeloid-derived cell populations | Up to 4 years
  The profile changes of the markers for immune cell activity, suppression, and exhaustion in T cell and myeloid-derived cell populations in response to ppDC assessed by cellular indexing of transcriptomes and epitopes-sequencing and a multi-color fluorescence-activated cell sorting panel.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony C Wang, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States